CLINICAL TRIAL: NCT06487754
Title: New-onset Chronic Pelvic Pain in Transgender People Using Testosterone Therapy: an Exploratory Qualitative Study.
Status: Recruiting | Type: Observational
Sponsor: University Hospital, Grenoble (Other)
Responsible Party: Sponsor
Other Study IDs: 24.01249.000416
Record Dates: First submitted 2024-06-19; First posted 2024-07-05 (Actual); Last update posted 2024-12-17 (Actual); Status verified 2024-12

CONDITIONS: Transgender Persons; Pelvic Pain; Testosterone; Gender-Affirming Care
MeSH Terms: conditions — Pelvic Pain

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
This descriptive qualitative study aim to describe the characteristics of pelvic pain in transgender (trans) individuals using testosterone therapy and the impact on their quality of life. This study also aim to understand the levers and obstacles to consulting a health care professional.

DETAILED DESCRIPTION:
This study ai to accurately describe the chronic pelvic plan (CPP) from which transmasculine people can suffer, as well as their impact on quality of life, and to understand what are the obstacles and levers to the implementation of adapted care.

Method: It is an observational, single-center, qualitative study. 10 to 15 trans individuals using testosterone therapy and having pelvic pain for at least 6 months, and that had appeared or changed since taking testosterone, will undergo a semi-structured interview. They will be recruited through community care associations, mailing lists and flyers.

Results: This is a qualitative study aimed at accurately describing the symptoms of pelvic pain experienced by trans people thus we will do a qualitative analysis. QCAMAPS will be used for the coding step.

ELIGIBILITY:
Inclusion Criteria:

* Being a trans masculine individual
* Taking a gender affirming hormonal therapy (GAHT)
* living close to Grenoble
* having pelvic pain that appeared or were modified after taking GAHT

Exclusion Criteria:

* Subject under guardianship or subject deprived of liberty Refusal of voice recording

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — trans masculine individual
Study Population: Trans masculine individuals using a gender affirming hormonal therapy (testosterone) and having pelvic pain.
Sampling Method: Non-Probability Sample
Enrollment: 15 (Estimated)
Dates: Start 2024-09-27 (Actual); Primary Completion 2025-02 (Estimated); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
Pelvic pain and impact on quality of life description | 1.5 hours during semi structured interviews
  Verbatim from the semi structured interviews

SECONDARY OUTCOMES:
pelvic pain intensity at the time of the interview | at the beginning of the interview
  visual analog scale from 0 to 100 mm

CONTACTS AND LOCATIONS:
Locations (1):
- UGA, Saint-Martin-d'Hères, France